CLINICAL TRIAL: NCT04553172
Title: Endothelial Dysfunction Leads to Bleeding Diathesis
Brief Title: Vascular Abnormalities and Bleeding Diathesis
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0471
Record Dates: First submitted 2020-09-02; First posted 2020-09-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2020-09

CONDITIONS: Bleeding Diathesis
Keywords: mucocutaneous bleeding; surgery bleeding outcomes
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected family members: Affected family members
- Affected PM: Affected PM

SUMMARY:
Inherited bleeding disorders (IBD) consist of a heterogeneous group of diseases including coagulation and/or platelets defects and more rarely vascular dysfunctions. A family of four patients suffering from unexplained excessive bleeding has been followed clinically in France for many years. Recently, whole exome sequencing (WES) of DNA allowed the identification of a heterozygous genetic variant which segregated to family members with bleeding diathesis. The aim of the study was to better characterize the phenotype by studying VWF and platelets in affected family members ultimately contributing to the pathogenesis of a bleeding diathesis.

DETAILED DESCRIPTION:
As explained in the brief summary, whole exome sequencing (WES) of DNA was performed in a family of four patients suffering from unexplained excessive bleeding. It allowed the identification of a variant which segregated to family members with bleeding diathesis. Firstly, in vitro, functional analyses were performed in primary human endothelial cells. Then, in-vivo analysis have to be performed on affected patients.

The four related patients suffering from excessive bleeding have been followed clinically in France for many years. During the follow-up of three of these affected patients, biological studies are planned.

Biological assays include:

* Conventional assessment of primary haemostasis: platelet count, platelet aggregation, functional and antigen measurement of von Willebrand factor.
* Specific testing: Von Willebrand factor multimeric profile, immunolabeling of platelets.

Conventional assessment is part of the conventional follow-up of patients with inherited bleeding disorder. It will not require any additional blood sample. For specific testing and after informed consent, fresh blood samples of patients will be collected in 1/10 volume of acid-citrate-dextrose and centrifuged for 10 min at 200 g to obtain Platelet-rich plasma (PRP) for functional analysis of platelets and Platelet-poor plasma for the multimerization state of von Willebrand factor. Then, the results will be compared to the in-vitro findings.

ELIGIBILITY:
Inclusion criteria:

- members of the family

Exclusion criteria:

- patient who refused to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A specific Family
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
platelet count | 1 day
  automatic count of platelet
platelet aggregation | 1 day
  automated assay using adenosine diphosphate (ADP), arachidonic acid (AA) agonists
VWF (von Willebrand factor) | 1 day
  activity/antigen levels measurements

SECONDARY OUTCOMES:
VWF mutimerization status | 1 day
  multimer distribution
immunostaining of platelets | 2 to 3 days
  fixed platelet studies coverslips are challenged with a panel of primary antibodies for immunofluorescence staining

CONTACTS AND LOCATIONS:
Overall Officials: Muriel GIANSILY-BLAIZOT, Principal Investigator — UH Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC